CLINICAL TRIAL: NCT06401746
Title: Assessment of Gastric Function Using Body Surface Gastric Mapping in Patients on Semaglutide (Ozempic)
Brief Title: Body Surface Gastric Mapping in Patients on Semaglutide
Status: Recruiting | Type: Observational
Sponsor: University of Western Sydney (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Vincent Ho, Associate Professor, University of Western Sydney
Other Study IDs: WS-GLP-001
Record Dates: First submitted 2024-04-28; First posted 2024-05-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Semaglutide-Induced Gastric Motility; Gastroparesis
Keywords: Semaglutide; GLP-1 Receptor Agonist; Gastric Motility; Body Surface Gastric Mapping
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Semaglutide: Patients undergoing Body Surface Gastric Mapping before and after administration of Semaglutide.
  Interventions: Device: Gastric Alimetry

INTERVENTIONS:
Device: Gastric Alimetry — The Gastric Alimetry™ System is intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of various gastric disorders.

SUMMARY:
Glucagon-like receptor-1 agonists (GLP-1 RAs), such as Semaglutide (Ozempic), are a class of drugs used for glycemic control in diabetes, and for weight loss and management in obesity. It has been shown to delay gastric emptying and lead to gastrointestinal symptoms. However, the exact mechanisms are unknown. Alterations in gastric function, including myoelectrical activity, may be a likely mechanism of gastrointestinal side effects.

Body Surface Gastric Mapping (BSGM) using the FDA-approved medical device Gastric Alimetry is a novel non-invasive diagnostic tool to assess gastric myoelectrical activity and patient-reported symptoms to achieve accurate non-invasive biomarkers of gastric dysfunction. A proof-of-principle case study of Ozempic using Gastric Alimetry showed abnormal gastric myoelectrical activity along with the development of severe bloating following the meal after 5 weeks of Ozempic use.

This study will extend on this initial finding by conducting an exploratory pilot study to investigate the effects on gastric motility in patients with and without diabetes before and after Ozempic. It is hypothesized that Gastric Alimetry will show changes in gastric myoelectrical activity and symptoms in patients after being on the weekly injectable Ozempic compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* No gastrointestinal symptoms based on Rome IV criteria
* For diabetics: Diagnosed T2DM (defined as HbA1c levels > 7%)
* For diabetics: Fasting blood glucose level < 15 mmol/L

Exclusion Criteria:

* Current use of Ozempic, similar GLP-1 RAs or regular insulin in the last 3 months
* Confirmed gastroparesis on gastric emptying scintigraphy
* Pregnant or breast-feeding
* Inability to perform a BSGM test according to Indications for Use: history of severe skin allergies or sensitivity to cosmetics or lotions; chronically damaged or vulnerable epigastric skin (fragile skin, wounds, inflammation); unable to remain in a relaxed reclined position for the test duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without Type 2 Diabetes Mellitus who are prescribed Semaglutide in a general metabolic clinic.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in overall postprandial BSGM Gastric Alimetry Rhythm Index (minimum: 0; maximum: 1) on treatment compared to baseline (with a lower score meaning worse outcome). | 3 months

SECONDARY OUTCOMES:
Change in Gastroparesis Cardinal Symptom Index (minimum: 0; maximum: 5) scores on treatment compared to baseline (with a higher score meaning worse outcome). | 3 months
Change in Patient Assessment of Upper Gastrointestinal Symptom Severity Index (minimum: 0; maximum: 5) scores on treatment compared to baseline (with a higher score meaning worse outcome). | 3 months
Change in Patient Assessment of Upper GastroIntestinal Disorders-Quality of Life (minimum: 0; maximum: 5) scores on treatment compared to baseline (with a lower score meaning worse outcome). | 3 months.
Change in 5-level EQ-5D (minimum: 0; maximum: 1) scores on treatment compared to baseline (with a lower score meaning worse outcome). | 3 months.
Change in Patient Health Questionnaire -8 (minimum: 0; maximum: 24) scores on treatment compared to baseline (with a higher score meaning worse outcome). | 3 months.
Change in General Anxiety Disorder-7 (minimum: 0; maximum: 21) scores on treatment compared to baseline (with a higher score meaning worse outcome). | 3 months.
Change in Perceived Stress Scale-4 (minimum: 0; maximum: 4) scores on treatment compared to baseline (with a higher score meaning worse outcome). | 3 months.
Correlation of postprandial BSGM Gastric Alimetry Rhythm Index (minimum: 0; maximum: 1) with symptom score (with a higher correlation meaning worse outcome). | 3 months.
  Symptoms scales are Gastroparesis Cardinal Symptom Index (minimum: 0; maximum: 5) and Patient Assessment of Upper Gastrointestinal Symptom Severity Index (minimum: 0; maximum: 5).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MBBS, FRACP, FACP, PhD, Principal Investigator — Western Sydney University
Locations (1):
- Western Sydney University, Campbelltown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kryger RA, Kolata JJ, Chung W, Dixit S, Tighe RJ, Vega JJ, DeYoung PA, Copi C, Sarafa J, Kovar DG, Gilfoyle GP, Sigworth SK. Two-particle correlations from neutron-light-charged-particle coincidences. Phys Rev Lett. 1990 Oct 22;65(17):2118-2121. doi: 10.1103/PhysRevLett.65.2118. No abstract available. PMID 10042458
- [Background] Wang WJ, Foong D, Calder S, Schamberg G, Varghese C, Tack J, Xu W, Daker C, Carson D, Waite S, Hayes T, Du P, Abell TL, Parkman HP, Huang IH, Fernandes V, Andrews CN, Gharibans AA, Ho V, O'Grady G. Gastric Alimetry Expands Patient Phenotyping in Gastroduodenal Disorders Compared with Gastric Emptying Scintigraphy. Am J Gastroenterol. 2024 Feb 1;119(2):331-341. doi: 10.14309/ajg.0000000000002528. Epub 2023 Oct 30. PMID 37782524
- [Background] Varghese C, Schamberg G, Calder S, Waite S, Carson D, Foong D, Wang WJ, Ho V, Woodhead J, Daker C, Xu W, Du P, Abell TL, Parkman HP, Tack J, Andrews CN, O'Grady G, Gharibans AA. Normative Values for Body Surface Gastric Mapping Evaluations of Gastric Motility Using Gastric Alimetry: Spectral Analysis. Am J Gastroenterol. 2023 Jun 1;118(6):1047-1057. doi: 10.14309/ajg.0000000000002077. Epub 2022 Dec 20. PMID 36534985